CLINICAL TRIAL: NCT02909036
Title: Pharmacokinetic (PK)-Directed Dosing of Captisol Enabled Melphalan for Patients With Multiple Myeloma or Light Chain (AL) Amyloidosis Undergoing High Dose Therapy and Autologous Hematopoietic Progenitor Cell Transplant
Brief Title: Study of Captisol Enabled Melphalan and Pharmacokinetics for Patients With Multiple Myeloma or Light Chain Amyloidosis That Are Receiving an Autologous Transplant.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-875
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma; Amyloidosis
Keywords: Melphalan; Autologous Hematopoietic Progenitor Cell Transplant; High Dose Therapy; 16-875
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis | interventions — pegfilgrastim

ARMS (1):
- Melphalan (Experimental): Test Dose CE Melphalan 10mg/m2 with PK studies Day -12 to Day-3, CE Melphalan Dose of Target AUC 13 mg/L/h infused with PK studies Day -2, 3-10 x 10^6 CD 34+ cells/kg reinfused Day 0, Pegfilgrastim 6mg injection Day +1
  Interventions: Device: Melphalan; Drug: Pegfilgrastim; Procedure: Autologous Hematopoietic Progenitor Cell Transplant

INTERVENTIONS:
Device: Melphalan
Drug: Pegfilgrastim
Procedure: Autologous Hematopoietic Progenitor Cell Transplant

SUMMARY:
Captisol Enabled Melphalan, is a new formulation of the standard of care melphalan chemotherapy that in packaged in an inactive substance that is believed to help the chemotherapy be more stable (meaning that it doesn't lose its effect or need to be administered quickly after being mixed). It may also have fewer side effects such as problems with important levels of body electrolytes such as potassium, phosphorous and magnesium; and cause less kidney and heart damage] than standard formulation melphalan.

The purpose of this study is to determine if the investigators can achieve a certain level of Captisol Enabled Melphalan that would be best to use in treating Multiple Myeloma and AL Amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 75
* Patients must have either:

  * Symptomatic multiple myeloma who have responded to prior induction or salvage chemotherapy (i.e. chemosensitive disease): Patients who are receiving high-dose melphalan and AHCT as part of their initial therapy require at least a partial response (PR) as defined by the International Myeloma Working Group uniform response criteria for MM.

Patients who are receiving high-dose melphalan and AHCT as part of salvage therapy require at least a minor response to their last line of therapy to document chemosensitive disease. There is no limit on the number of prior regimens received by the patient.

OR

* Light chain (AL) amyloidosis who may be newly diagnosed or previously treated

  * Histologic and serologic findings, reviewed at MSKCC, confirming the diagnosis of multiple myeloma or AL amyloidosis. Standard diagnostic criteria for multiple myeloma will be used, as per the International Myeloma Foundation consensus guidelines
  * Patients must have at least 3 x 10^6 CD34+ cells/kg frozen.
  * Adequate organ function is required, defined as follows:
* Serum bilirubin ≤ 2.0 mg/dl
* AST, ALT and alkaline phosphatase < 3 times the upper limit of laboratory normal
* Creatinine clearance ≥ 40 ml/min (24 hour urine collection)
* LVEF ≥ 45% by MUGA or rest ECHO
* Diffusing capacity ≥ 45% (adjusted for hemoglobin) predicted by pulmonary function testing
* Performance status (ECOG) ≤ 2

  * A willingness to avoid pregnancy or fathering children in male and female subjects respectively
* A woman of childbearing potential must have a negative serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at screening and must be willing to avoid pregnancy during the study treatment period and for a specified duration (1 year post HCT) after the end of treatment.
* Women of childbearing potential who have a negative serum pregnancy test at screening must practice a highly effective method of birth control (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the subject and their understanding confirmed.
* Men who are enrolled must agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the subject and their understanding confirmed

Exclusion Criteria:

* Unstable angina or myocardial infarction within 4 months of initiating therapy on trial, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
* Light chain (AL) amyloidosis patients with Mayo Cardiac Stage IIIB (defined as NT-proBNP>8500 ng/L and Cardiac troponin (cTnT) >0.035 μg/L)
* Pregnant or lactating females
* Nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Contraindication to CE melphalan or any of the required supportive treatments, including hypersensitivity to G-CSF or pegfilgrastim
* Any other medical condition or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial
* Any known allergy or allergic reactions to Captisol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 day
  defined as stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR) to high-dose CE melphalan in patients enrolled in the study between days 90-100 post-AHCT. Responses will be evaluated by the IMWG Response Criteria and Minor Response (MR) criteria. Responses will be evaluated by the standard AL Amyloid Organ Response Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/